CLINICAL TRIAL: NCT06656923
Title: PLLA-ADIPOGENESIS-IFA: Immunofluorescence Analysis to Quantify Changes Induced by Poly-L-Lactic Acid in Adipose Tissue
Brief Title: Analyze Previously Collected Biopsy Samples From Participants Who Completed the "SPLASH: Split-Body Randomized Clinical Trial of Poly-L-Lactic Acid for Adipogenesis and Volumization of the Hip Dell" Study
Status: Active, not recruiting | Type: Observational
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: PLLA-HIP-DELL-STAINS-2024
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-10

CONDITIONS: Lateral Gluteal Depression
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Biopsies — Analyze previous biopsies to quantify changes induced by Poly-L-Lactic Acid in Adipose Tissue

SUMMARY:
Primary Objective: use immunofluorescence (IF) on previously obtained biopsies to analyze and quantify changes in adipose tissue of subjects injected with poly-L-lactic acid (PLLA) or saline.

DETAILED DESCRIPTION:
Sixteen female adults that participated in SPLASH study will be enrolled in this retrospective study. It aims to analyze previously collected biopsy samples from participants who completed the "SPLASH: Split-Body Randomized Clinical Trial of Poly-L-Lactic Acid for Adipogenesis and Volumization of the Hip Dell" study. The study will use immunohistology to assess changes in adipose tissue associated with treatment with PLLA (poly-L-lactic acid). We hypothesize that specimens treated with PLLA will be found to have more adipocyte-derived stem cells and preadipocytes undergoing mitosis and differentiation compared to control specimens.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed all biopsies in the previous SPLASH trial "A Single Center, Double- Blinded, Split-Body, Randomized Clinical Trial of Injectable Poly-L-Lactic Acid for Volumization and Adipogenesis of the Hip Dell - Protocol Number Sculptra-Hip-Dell-2021-12" .

Exclusion Criteria:

* Subjects who had biopsies of poor quality, insufficient tissue, or were otherwise unsuitable for immunofluorescence analysis.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Previous study was only done on females due to skin quality and aesthetic concerns
Study Population: 16 Females that were previously enrolled and biopsied in SPLASH study.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in cell count per area between PLLA and saline-treated specimens. | Specimens are from 6 months post-treatment compared to pre-treatment / Baseline
  Analyzing between PLLA and saline-treated specimens for the following populations:
  * adipocyte derived stem cells
  * proliferating adipocyte-derived stem cells
  * preadipocytes/adipocyte precursors
  * proliferating preadipocytes/adipocyte precursors
  * mature adipocytes and actively differentiating precursors The following proteins will be quantified and the differences between PLLA and saline-treated specimens at 6 months compared to pre-treatment will also be analyzed:
  * β-catenin
  * PPARγ
  * Adiponectin
  * Perilipin-1

CONTACTS AND LOCATIONS:
Locations (1):
- Cosmetic Laser Dermatology/West Dermatology Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No